CLINICAL TRIAL: NCT04154618
Title: Continuous Vital Sign Monitoring in Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Barry Weinberger, Principal Investigator, Northwell Health
Other Study IDs: 19-0653
Record Dates: First submitted 2019-10-11; First posted 2019-11-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Newborn Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous wireless vital sign monitoring — Infants will receive wireless vital sign monitoring throughout their birth hospitalization.

SUMMARY:
This study evaluates the feasibility and usability of continuous wireless vital sign monitoring of well newborns during their birth hospitalization.

DETAILED DESCRIPTION:
This study is conducted for the purposes of understanding the feasibility and acceptability of routine wireless continuous monitoring on healthy newborns as a standard practice & its effect on existing workflows and as a future tool for the early detection of undiagnosed problems. All infants will receive routine newborn nursing care .

Once alarm limits have been determined, the monitoring data will be analyzed in real time and out of range vital signs will alert the nurse to perform standard assessment of the newborn.

Nurse and parents will complete surveys regarding their experience with continuous vital sign monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants <12 hours of age
* Expected to be admitted to the Well Baby Nursery
* 36 or more weeks gestation at birth
* Mother at least 18 years of age

Exclusion Criteria:

* Infants requiring any non-routine medical care or observation
* Neonatal Intensive Care Unit (NICU) or Special Care Nursery admission
* Multiple birth

Ages: 0 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy newborn infants < 12 hours of age admitted to the Well Baby Nursery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of feasibility by questionnaires to nurses and mothers using the using the Technology Acceptance Model (TAM). | Up to 3 days
  TAM questionnaires will be distributed to the nurse taking care of each subject at the time of discharge of the infant. The questionnaire will include informed consent by the nurse for participation in the research. A similar questionnaire will also be distributed to the mother just prior to discharge.

SECONDARY OUTCOMES:
Accuracy assessed by comparison to conventional vital sign measurements within a 2-minute window | Up to 3 days
  The mean continuous measurements within a 2-minute window around each conventional vital sign assessment (routinely, several in the first 4 hours after birth, and then every 12 hours) will be compared to the routine measurement.
Clinical Utility as measured by false alerts | Up to 3 days
  Quantify false positive alerts and false negative alerts as a measure of potential adverse effect on nursing workflow and patient care

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Phelps Hospital, Sleepy Hollow, New York

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD).
Supporting Information: CSR
Time Frame: Data will become available after enrollment is complete and all data have been collected
Access Criteria: Requests to the principal investigator (PI) to obtain data outlining the purpose of the study, the data elements to be accessed, preferred method of transmission, and preferred file type. For requests of identifiable information or information utilizing a limited data set a copy of valid institutional review board (IRB) approval and informed consent, as applicable. The PI will evaluate the request and ensure that appropriate regulatory approvals have been obtained. Once approved the investigator will be informed and relevant data transferred for analysis.